CLINICAL TRIAL: NCT00033839
Title: A Phase III, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multicenter Evaluation of Civamide (Zucapsaicin) Nasal Solution in the Treatment of Episodic Cluster Headache
Brief Title: A Phase III Study of Civamide Nasal Solution (Zucapsaicin) for the Treatment of Episodic Cluster Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Winston Laboratories (Industry)
Responsible Party: Scott B. Phillips, M.D., Study Director, Winston Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WL-1001-02-02
Record Dates: First submitted 2002-04-11; First posted 2002-04-12 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Episodic Cluster Headache
Keywords: Headache; Cluster; EC; Episodic Cluster
MeSH Terms: conditions — Cluster Headache; Headache | interventions — zucapsaicin

INTERVENTIONS:
Drug: Civamide (Zucapsaicin)

SUMMARY:
This is a 49-day study to evaluate the effectiveness of Intranasal Civamide (Zucapsaicin) in the treatment of an episodic cluster headache period compared to placebo (medically inactive substance which does not contain any active ingredients).

ELIGIBILITY:
* At least 2 year history of episodic cluster headache (meeting IHS criteria)
* At least 2 previous episodes
* Expected duration of cluster period is at least 6 weeks but not longer than 16 weeks
* At least 1 but not more than 8 headaches on each of the 3 days immediately prior to treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-01; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott B. Phillips, M.D., Study Director — Winston Laboratories
Locations (26):
- United States (26):
  - Valley Neurological Headache & Research Center, Phoenix, Arizona
  - Neurological Associates of Tucson, Tucson, Arizona
  - Northern California Headache Clinic, Mountain View, California
  - San Francisco Clinical Research Center, San Francisco, California
  - California Medical Clinic for Headache, Santa Monica, California
  - New England Center for Headache, PC, Stamford, Connecticut
  - Neurology Clinical Research, Inc., Plantation, Florida
  - Neurology and Headache Specialists of Atlanta, Decatur, Georgia
  - Diamond Headache Clinic, Chicago, Illinois
  - Boston Clinical Research Center, Wellesley Hills, Massachusetts
  - Michigan Headache Pain & Neurological Institute, Ann Arbor, Michigan
  - Henry Ford Hospital Department of Neurology, Detroit, Michigan
  - Department of Neurology Mayo Clinic, Rochester, Minnesota
  - Mercy Health Research, Chesterfield, Missouri
  - Headache Care Center/Clinvest, Springfield, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - New York Headache Center, New York, New York
  - The Headache Wellness Center, Greensboro, North Carolina
  - Cincinnati Headache Clinic, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Neurological Associates of Tulsa, Inc., Tulsa, Oklahoma
  - Jefferson Headache Center, Philadelphia, Pennsylvania
  - Nashville Neuroscience Center, Nashville, Tennessee
  - Houston Headache Clinic, Houston, Texas
  - The Neurology and Headache Treatment Center (Innovative Clinical Research), Alexandria, Virginia